CLINICAL TRIAL: NCT06278649
Title: Relaxation and Guided Imagery as an Intervention for Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pace University (Other)
Collaborators: University of Connecticut (Other); Touro University (Other)
Responsible Party: Principal Investigator, Johanna deLeyer-Tiarks, Assistant Professor, Pace University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-161-Multi-site
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Anxiety
MeSH Terms: conditions — Asthma; Anxiety Disorders | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relaxation and Guided Imagery Intervention (Experimental): During the RGI sessions, the participant will be told to lie down on an exercise mat while a 15 minute relaxation and guided imagery audio recording is played. During the relaxation portion of the script, the participant will be instructed to let go of tension they might feel in individual parts of their body (starting with their feet and working their way up). The second portion is the guided imagery portion, which includes asking each participant to imagine themselves in a peaceful place. The participant will then be guided to imagine healing in the specific bronchial tubes and lungs, asking them to imagine themselves doing a favorite activity in which they have no trouble with their asthma, and asking them to visualize breathing in a colored air that would clear the airways and lungs.
  Interventions: Behavioral: Relaxation and Guided Imagery

INTERVENTIONS:
Behavioral: Relaxation and Guided Imagery — Listening to a 15 minute relaxing pre-recorded script while laying down on an exercise mat

SUMMARY:
The purpose of the current study is to investigate the usefulness of a Relaxation and Guided Imagery intervention for the reduction of asthmatic symptoms in adults and children whose asthma symptoms are aggravated, or triggered by anxiety. This study will replicate the previous literature to further investigate the impact that a Relaxation and Guided Imagery intervention can have on anxiety and related asthmatic symptoms using a multiple baseline (small sample size) research design. Participants will fill out questionnaires, listen to RGI audio tapes, and provide lung functioning samples by blowing into a spirometer.

DETAILED DESCRIPTION:
The purpose of the current study is to investigate the usefulness of a Relaxation and Guided Imagery intervention for the reduction of asthmatic symptoms in individuals whose asthma symptoms are aggravated, or triggered by anxiety. Relaxation and Guided Imagery (RGI) techniques have been used to assist in the reduction of anxiety symptoms in several experimental studies. Various psychologically-based treatments have been effective in treating asthmatic symptoms. This study will replicate the previous literature to further investigate the impact that a Relaxation and Guided Imagery intervention can have on anxiety and related asthmatic symptoms.

Research Questions and Hypotheses:

1. Will a Relaxation and Guided Imagery intervention reduce asthma symptoms?

1a. It is hypothesized that an RGI intervention will reduce participants' asthma symptoms from pre-intervention to post-intervention as measured by Forced Vital Capacity (FVC) & Forced Expiratory Airflow (FEV).

2. Will a Relaxation and Guided Imagery intervention reduce anxiety?

2a. It is hypothesized that an RGI intervention will reduce participants' anxiety from pre-intervention to post-intervention as measured by the State-Trait Anxiety Inventory.

3. Will a Relaxation and Guided Imagery intervention increase quality of life?

3a. It is hypothesized that an RGI intervention will increase participants' quality of life from pre-intervention to post-intervention as measured by the Asthma Quality of Life Questionnaire (AQLQ).

Design: This study will utilize a multiple-baseline research design with three to five participants. Three participants are sufficient to demonstrate a functional relationship between the intervention and the outcome measure; however, additional participants may be included to strengthen the case and provide some protection from attrition. With this design, we will be able to show three demonstrations of change at three different points in time, which is a widely accepted convention in the field of single-subject research for demonstrating a functional relationship between the independent variable and the outcome measures.

Recruitment → Screening → Intake → Baseline → Intervention → Post Treatment → Maintenance

Recruitment. Participants will be recruited from the community. Specifically, the study will be advertised through web-based communication platforms (e.g. newsletters, listservs, community forums) and printed flyers (see attached recruitment materials). There will be no compensation or "bonuses" for participant recruitment.

Screening. All screening procedures will take place through videoconferencing, or in the PIs' office either on the Pace University campus or University of Connecticut Campus. Prospective participants who consent to the screening (see attached Screening Consent forms) will be asked to complete the following procedures: (1) an interview to gather the inclusionary and exclusionary information, and (2) the Trait Form of the State-Trait Anxiety Inventory (or, for prospective child participants, the Trait form of the State-Trait Anxiety Inventory for Children). Prospective participants (or, for prospective child participants, their legal guardians) will be notified via email with the screening result, and those who have met screening criteria for inclusion will be asked to schedule a time to complete an intake meeting (see attached email script). Any data collected from individuals who do not meet inclusionary criteria will be destroyed immediately.

Intake. All intake procedures will take place in the PIs' office either on the Pace University campus or University of Connecticut Campus. In an intake meeting, the purposes and activities of the study will be explained to prospective participants and/or their legal guardians. Following this, adults will be given a consent form to review for signature and given time to answer questions (see attached Consent Form). For children/adolescents, assent will be obtained (see attached Child Assent Script) and legal guardians will be given a permission form to review for signature and given time to answer questions (see attached Permission Form). Once consent (or, for child participants, permission) is obtained, participants will be asked to provide a forced vital capacity (FVC) and forced expiratory air-flow (FEV1) reading using a calibrated spirometer, complete the Asthma Quality of Life Questionnaire (AQLQ), (or, for child participants, the Pediatric Asthma Quality of Life Questionnaire (PAQLQ)).

Baseline. During the baseline phase, data on each participant will be collected once weekly for approximately four weeks in a PIs office on the following measures: (1) State form of the STAI (or, for child participants, the STAIC), (2) FEV1 and FVC, and (3) Daily Asthma Logs. Each baseline phase session will last for approximately 30 minutes. The RGI intervention will not be implemented during this phase.

Intervention. During the intervention phase the Relaxation and Guided Imagery (RGI) intervention will be implemented. Data on each participant will be collected once weekly for approximately four weeks in a PIs office on the following measures: (1) State form of the STAI (or, for child participants the STAIC), (2) FEV1 and FVC, and (3) Daily Asthma Logs (see attached Daily Asthma Log). Each intervention phase session will last for approximately 1 hour. Participants will complete intervention phase activities in the following order: (1) fill out the STAI or STAIC, (2) provide an FEV1 and FVC reading, (3) complete the RGI intervention (see below), (4) provide a second FEV1 and FVC, and (5) fill out the STAI or STAIC again.

Relaxation and Guided Imagery Intervention. During the RGI sessions, the participant will be told to lie down on an exercise mat while a 15 minute relaxation and guided imagery audio recording is played. During the relaxation portion of the script, the participant will be instructed to let go of tension they might feel in individual parts of their body (starting with their feet and working their way up). The second portion is the guided imagery portion, which includes asking each participant to imagine themselves in a peaceful place. The participant will then be guided to imagine healing in the specific bronchial tubes and lungs, asking them to imagine themselves doing a favorite activity in which they have no trouble with their asthma, and asking them to visualize breathing in a colored air that would clear the airways and lungs.

Post Treatment. Following the intervention phase, participants will meet with the researchers in a PIs' office to complete the same measures that were given during the pre-test and baseline phases. This includes both the State and Trait forms of the STAI (or, for child participants, the STAIC), the AQLQ (or, for child participants, the PAQLQ), FVC and FEV1. Participants will also be asked to complete the Consumer Satisfaction Questionnaire- Revised (CSQ-R).

Maintenance. During this phase, two follow ups will occur, one short-term follow up at four weeks post-intervention and one long-term follow up at three months post-intervention. The study team will contact participants via email (see attached email scripts) and ask that they attend a meeting to complete the follow-up measures. The follow-up measures, for both short- and long-term, include the State and Trait forms of the STAI (or the STAIC for child participants), FVC and FEV1, and the AQLQ (or the PAQLQ for child participants). Following this, participants will be given copies of the RGI intervention audio recording which can be practiced independently after the conclusion of the study.

Duration

Screening: One approximately 45 minute meeting (Total time: ~45 min)

Intake: One approximately 30 minute meeting (Total time: ~30 min)

Baseline Phase: Once weekly approximately 30 minute meetings over 3-5 weeks (Total time: ~1.5 hours - ~2.5 hours)

Intervention Phase: Once weekly approximately 1 hour minute meetings over 3-5 weeks (Total time: ~3 hours - ~5 hours)

Post Treatment Phase: One approximately 45 minute meeting (Total time: ~45 min)

Maintenance Phase: Two approximately 30 minute meetings occurring at one month and three months post-program. (Total time: ~1 hours)

ELIGIBILITY:
Inclusion Criteria:

* At least 8 years of age and no older than 80 years of age
* Have clinical levels of anxiety
* Report having asthma
* Have asthma symptoms become triggered or exacerbated by anxiety

Exclusion Criteria:

* Under 8 years old or older than 80 years old
* No clinical levels of anxiety
* No asthma symptoms triggered or exacerbated by anxiety

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Asthma | Taken during weekly meeting occuring for 3-5 weeks during pre-intervention period, 3-5 weeks during intervention period, 1 week during the post-intervention period
  Lung functioning as measured through spirometry data (Forced Vital Capacity)
Asthma | Taken during weekly meeting occuring for 3-5 weeks during pre-intervention period, 3-5 weeks during intervention period, 1 week during the post-intervention period
  Lung functioning as measured through spirometry data (Forced Expiratory Volume 1)
Anxiety | Taken during weekly meeting occuring for 3-5 weeks during pre-intervention period, 3-5 weeks during intervention period, 1 week during the post-intervention period
  Anxiety as measured by the State-Trait Anxiety Inventory; measures general levels of anxiety (trait) and current levels of anxiety (state) on a scale from 20 (minimum) to 80 (maximum) with higher scores corresponding to higher levels of anxiety (lower score = better outcome)

SECONDARY OUTCOMES:
Quality of Life | Taken during one pre-intervention meeting and one post-intervention
  Quality of life as measured by the Asthma Quality of Life Questionnaire; measures physical and emotional quality of life, including symptoms, emotional function, and limitations engaging in daily activities on a scale from 32 (minimum) to 224 (maximum) with lower scores corresponding to higher levels of quality of life (lower score = better outcome).

IPD SHARING:
Plan to Share IPD: No